CLINICAL TRIAL: NCT00955864
Title: Non-Invasive Non-Ionizing Polarized Imaging System to Assess Structure of Cervix
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090180; 09-CH-0180
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-09-01

CONDITIONS: Healthy
Keywords: Cervix; Colposcope; Polarized Light; Cervix Structure; Collagen; HV; Healthy Volunteer; Healthy Women

SUMMARY:
Background:

* The uterine cervix is composed of muscle and collagen, which change as women age and under hormonal influences like puberty, pregnancy, and menopause. Yet even though knowledge of structure of the cervix (especially the collagen network) is important to detect problems that may affect pregnancy and other women s health issues, no noninvasive techniques are available to evaluate such changes.
* A specially designed polarized camera attached to a conventional colposcope can be used to take cervical images. Analyzing these images may enable researchers to better visualize the collagen network in the cervix.

Objectives:

* To explore and gain experience with the use of a polarized imaging system to study cervical structure.
* To evaluate the usefulness of a polarized imaging system in studying the cervical structure of healthy nonpregnant women.

Eligibility:

- Adult females (at least 18 years of age) who are having regular menstrual cycles and are not on hormonal medications.

Design:

* Images will be takes from the cervix in two different phases of menstruation cycle time, one in the follicular phase (before ovulation) and another one in the luteal phase (after ovulation).
* The images of the cervix will be taken with a vaginal speculum in place with the camera attached to a colposcope. The colposcope will illuminate the cervix using polarized light. Three random cervical locations will be photographed

DETAILED DESCRIPTION:
The uterine cervix is composed of muscle and collagen which changes as women age and under hormonal influences like after puberty, during pregnancy, and with menopause. It has been determined that during pregnancy, prior to cervical ripening, cross linked collagen fibrils are organized in tight bundles which provide tensile strength, rigidity and stiffness. As the cervix ripens in preparation for labor, cervical collagen concentration is decreases and solubility increases. However, there are no noninvasive techniques available to evaluate such structural changes especially of the collagen of cervix. Developing a non-invasive way to evaluate the characteristics of cervical structure and collagen may aid in identifying women who are at risk of early cervical dilation. A specially designed polarized camera attached to a conventional colposcope can be used to take cervical images. Analyzing these images may enable us to visualize the collagen network in cervix. The purpose of this study is to explore the usefulness of polarized camera images in evaluating the cervical structure of healthy women at different ages. After evaluating and validating this approach in healthy, nonpregnant women, we plan to assess the cervical structure of pregnant women, some of whom may be at risk of early cervical dilation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age female 18 year or greater including IUI patients. Healthy women without significant medical problems who have a uterine cervix.

EXCLUSION CRITERIA:

* Those with symptoms or signs of infection or are currently menstruating.
* Any medical condition that, in the opinion of Principal Investigator, would preclude the inclusion of a patient onto this research study.
* Unable or unwilling to give informed consent.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07-15; Study Completion 2016-09-01

CONTACTS AND LOCATIONS:
Overall Officials: Amir Gandjbakhche, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Maul H, Mackay L, Garfield RE. Cervical ripening: biochemical, molecular, and clinical considerations. Clin Obstet Gynecol. 2006 Sep;49(3):551-63. doi: 10.1097/00003081-200609000-00015. PMID 16885662
- [Background] KRANTZ KE, PHILLIPS WP. Anatomy of the human uterine cervix, gross and microscopic. Ann N Y Acad Sci. 1962 Sep 29;97:551-63. doi: 10.1111/j.1749-6632.1962.tb34666.x. No abstract available. PMID 14035478
- [Background] Jacques SL, Roman JR, Lee K. Imaging superficial tissues with polarized light. Lasers Surg Med. 2000;26(2):119-29. doi: 10.1002/(sici)1096-9101(2000)26:23.0.co;2-y. PMID 10685085